CLINICAL TRIAL: NCT05387486
Title: Internal Jugular Vein Cannulation: A Comparison Of Three Techniques: Anatomical Landmark, US Guided Prelocation, and Ultrasound Guided Real Time, at Tertiary Care Teaching University Hospital
Brief Title: Central Venous Catheter Insertion Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Syed Shabbir Ahmed, Senior Instructor, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3488-Ane-ERC-15
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Catheterization, Central Venous
Keywords: Cardiac Surgery; Central Venous Catheter; Anatomical Landmark; Ultrasound

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ALT (Active Comparator)
  Interventions: Procedure: Anatomical Landmark technique
- USG-Pre (Active Comparator)
  Interventions: Procedure: Ultrasound-guided pre location technique
- USG -RT (Active Comparator)
  Interventions: Procedure: Ultrasound-guided real-time technique

INTERVENTIONS:
Procedure: Anatomical Landmark technique — anatomical landmarks (sternocleidomastoid muscles, sternal notch, cricoid cartilage, carotid artery and clavicle) will be palpated. A 3cc syringe with 21 gauge needle (locator) will be used first to locate IJV at the apex of the triangle formed by the two heads of the sternocleidomastoid muscle. After successful location, an introducer needle of 18 gauge, attached with a 5 ml syringe, will be inserted at the same point. The introducer needle will be directed towards the ipsilateral nipple at an angle of 20-30° with the skin
  Arms: ALT
Procedure: Ultrasound-guided pre location technique — In Group Ultrasound-guided pre location technique, venipuncture site will be determined using ultrasound probe which will be then removed and locator needle of 21 gauge will be used first to confirm IJV location. The cannulation or venipuncture will be performed at the marked point of locator needle by the use of 18 gauge introducer needle.
  Arms: USG-Pre
Procedure: Ultrasound-guided real-time technique — In Group Ultrasound-guided real-time technique, cannulation or venipuncture will be performed under real-time imaging using 18 gauge needle i-e ultrasound will be used for prelocation and puncturing of IJV and locator needle will not be used
  Arms: USG -RT

SUMMARY:
Investigator compared three techniques of Central venous cannulation (CVC) insertion, Anatomical Landmark, Pre-location Ultrasound and the Real Ultrasound techniques, in cardiac surgical patients.

DETAILED DESCRIPTION:
Central venous cannulation (CVC) is the cannulation of a large central vein in neck (internal jugular vein), chest (subclavian or axillary) or groin (femoral vein). It is a standard clinical method performed for the monitoring of central venous pressure, temporary haemodialysis, drug administration (drugs irritating peripheral veins, chemotherapy, concentrated vasoactive drugs ) rapid infusion of fluids, inadequate peripheral intravenous access and sampling site for repeated blood sampling. There are different techniques for Central venous cannulation which include anatomical landmark and ultrasound guided (USG) technique.

Previous studies have shown that the successful IJV cannulation using anatomical landmark technique was 85% as compared to ultrasound guided IJV cannulation which was 95%.The median catheterisation time of internal jugular vein via ultrasound guided (USG) is shorter than anatomical landmark technique.

There has been little evidence regarding the use of ultrasound guidance for internal jugular vein cannulation at a tertiary care hospital in our population. Furthermore with widespread availability of ultrasound, Internal Jugular vein can be successfully cannulated with decreasing number of attempts, less time consumption and decrease in the incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA (American society of Anesthesiologists) status 1 to 3 requiring central venous catheter during surgical procedure
* ASA (American society of Anesthesiologists) status 4 patients coming for cardiac surgery

Exclusion Criteria:

Patients with a history of following

* Previous head and neck surgery
* Head and neck mass or cancer.
* Superior vena cava syndrome.
* Coagulopathy.
* Infection at the cannulation site.
* Previous central venous access.
* Anatomical Changes due to surgery or any pathology in the neck which can lead to distortion of anatomical land marks in the region of puncture.
* Raised intracranial pressure (ICP).
* Patients coming for emergency surgery
* Patients with BMI (Body Mass Index) more than 30
* Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
Success Rate | Day 1
  Success rate will be measured according to the number of attempts. The cannulation of right Internal Jugular Vein within the first three attempts.

SECONDARY OUTCOMES:
Time duration for each technique | Day 1
  Measurment of time in minutes
Incidence of Complications | Day 1
  Look for carotid puncture, haematoma formation , pneumothorax

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ray BR, Mohan VK, Kashyap L, Shende D, Darlong VM, Pandey RK. Internal jugular vein cannulation: A comparison of three techniques. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):367-71. doi: 10.4103/0970-9185.117115. PMID 24106363
- [Background] Leung J, Duffy M, Finckh A. Real-time ultrasonographically-guided internal jugular vein catheterization in the emergency department increases success rates and reduces complications: a randomized, prospective study. Ann Emerg Med. 2006 Nov;48(5):540-7. doi: 10.1016/j.annemergmed.2006.01.011. Epub 2006 Feb 21. PMID 17052555
- [Background] Kaye AD, Fox CJ, Hymel BJ, Gayle JA, Hawney HA, Bawcom BA, Cotter TD. The importance of training for ultrasound guidance in central vein catheterization. Middle East J Anaesthesiol. 2011 Feb;21(1):61-6. PMID 21991734